CLINICAL TRIAL: NCT02998021
Title: Effect of Vibration Exercise on Upper Limb Strength, Function, and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alicia Koontz (Other)
Responsible Party: Sponsor-Investigator, Alicia Koontz, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO16010169
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Resistance Training - Vibrating Dumbbell (Experimental): Study participants who are randomized into the vibration exercise group will complete an in-home exercise program using a vibrating dumbbell.
  Interventions: Device: Vibrating Dumbbell
- Resistance Training - Standard Dumbbell (Active Comparator): Study participants who are randomized into the control exercise group will complete an in-home exercise program using standard dumbbells.
  Interventions: Device: Standard Dumbbell

INTERVENTIONS:
Device: Vibrating Dumbbell — Supervised training sessions will occur optimally, 3 times per week for a total of 12 consecutive weeks. The sessions will involve nine exercises specifically designed to improve upper limb muscle function. The beginning training intensity for each participant will be based on their one rep max for each exercise, which is determined during baseline laboratory testing in accordance with standard procedures. Training intensity will be adjusted progressively, first by increasing the frequency of the vibration (max. 40 Hz) then by the addition of more weight, based on weekly assessments and consultation with the senior investigators.
  Arms: Resistance Training - Vibrating Dumbbell
Device: Standard Dumbbell — Supervised training sessions will occur optimally, 3 times per week for a total of 12 consecutive weeks.
  The sessions will involve nine exercises specifically designed to improve upper limb muscle function. The beginning training intensity for each participant will be based on their one rep max for each exercise, which is determined during baseline laboratory testing in accordance with standard procedures. Training intensity will be adjusted progressively by the addition of more weight, based on weekly assessments and consultation with the senior investigators.
  To obtain as much data as possible on resistance training with vibration within study timeline, a modification was recently approved by the Institutional Review Board (IRB) to cease enrolling subjects into standard dumbbell training.
  Arms: Resistance Training - Standard Dumbbell

SUMMARY:
The primary purpose of this study is to explore the benefits of vibration dumbbell resistance training over standard dumbbell resistance training for improving upper limb strength, function and pain among manual wheelchair users with paraplegia.

DETAILED DESCRIPTION:
Objectives: The primary purpose of this study is to explore the benefits of vibration dumbbell resistance training over standard dumbbell resistance training for improving upper limb strength, function and pain among manual wheelchair users with paraplegia.

Experimental Design: Design: Randomized Control Trial

Methods: Twenty subjects with paraplegia will be recruited and randomized into two groups, a vibration dumbbell training (V-DT) group and a standard dumbbell training group (S-DT). Both groups will participate in a supervised 12-week (3 sessions per week) dumbbell (free-weight) strength training program consisting of nine exercises specifically designed to improve upper limb muscle function to support propulsion and transfer activities and protect the shoulders from developing pain. For each of the nine exercises the vibration group will hold a high-frequency (40 Hz) vibrating dumbbell in a static arm posture (isometric training) while the control group will move a non-vibrating dumbbell through the full range of motion for a given exercise (isotonic training). Both groups will follow a standardized protocol for assessing and progressing the amount of weight that is added to the dumbbell to achieve optimal training effects.

All participants will participate in laboratory testing for various outcome measures at baseline, 6 weeks and 12 weeks .

ELIGIBILITY:
Inclusion Criteria:

* have a neurological impairment secondary to spinal cord injury (SCI) or disease at T2 or lower
* greater than 6 months post injury
* use a manual wheelchair as primary means of mobility (at least 30 hrs. per week)
* 18 to 65 years of age
* provide signed medical release by primary care physician to engage in a high-intensity resistance training exercise program
* live within 60 minutes driving time (1 hour) from the research center
* able to perform a transfer independently to and from a wheelchair
* have normal range of motion in the upper limbs.

Exclusion Criteria:

* history of fractures or dislocations in the shoulder, elbow and wrist from which the subject has not fully recovered or joint replacement of any of the joints in the upper extremities
* upper limb pain that interferes with the ability to propel or transfer
* recent hospitalization for any reason (within the past three months)
* pregnant women
* history of coronary artery disease, coronary bypass surgery or other cardio-respiratory events

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Koontz, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Resistance Training - Standard Dumbbell: Study participants who are randomized into the control exercise group will complete an in-home exercise program using standard dumbbells.
  Standard Dumbbell: Supervised training sessions will occur optimally, 3 times per week for a total of 12 consecutive weeks.
  The sessions will involve nine exercises specifically designed to improve upper limb muscle function. The beginning training intensity for each participant will be based on their one rep max for each exercise, which is determined during baseline laboratory testing in accordance with standard procedures. Training intensity will be adjusted progressively by the addition of more weight, based on weekly assessments and consultation with the senior investigators.
  To obtain as much data as possible on resistance training with vibration within study timeline, a modification was recently approved by the IRB to cease enrolling subjects into standard dumbbell training.
Period: Overall Study
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Started | 8 | 2
Completed | 5 | 0
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — unsafe home | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.9) | 41.4 (3.5) | 46.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 1 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Strength
Description: Measurement of peak torque (Nm/kg) for Shoulder Adduction. Measurement was done using the Biodex System.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit. There were technical problems with collected the strength data for one subject in the intervention group.
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 4 | 0
Nm/kg | -4.0 (12.4) |

2. Primary Outcome: Change in Upper Extremity Pain
Description: Score generated by the Numerical Rating Scale for shoulder pain. Participants self report upper extremity pain over the last 24 hours with scores on a 0 to 10 scale. Higher scores represent higher levels of pain.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit
Measure: Median (Full Range); unit: units on the scale
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 5 | 0
units on the scale | 0 [-1 to 0] |

3. Primary Outcome: Change in General Health Measures
Description: Score generated by the Short Form 36 walk-wheel. Participants self report on health questions within 8 domains each of which are scored from 0 to 100. The scores from each of the subscales are then averaged together to obtain an overall total score. A score of 0 represents the worst possible health state and a score of 100 represents the best possible health state.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit
Measure: Mean (Standard Deviation); unit: units on the scale
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 5 | 0
units on the scale | 5.0 (15.3) |

4. Primary Outcome: Changes in Functional Shoulder Pain
Description: Score generated by the Wheelchair Users Shoulder Pain Index. Participants self report shoulder pain over the past week while performing activities of daily living. Scores range from 1 to 150 where higher scores represent higher levels of pain.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit
Measure: Mean (Standard Deviation); unit: units on the scale
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 5 | 0
units on the scale | 1.4 (10.2) |

5. Secondary Outcome: Change in Peak Speed
Description: Change in peak speed (m/s) measured on a 3 degree incline. Measurement will be done using the SmartWheel.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit. There were technical issues that prevented SmartWheel data collection for 3 subjects in the intervention group.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 2 | 0
meters/second | -0.08 (0.07) |

6. Secondary Outcome: Change in Acceleration
Description: Change in acceleration (seconds) during the 250 foot level propulsion task.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 5 | 0
seconds | 1.8 (2.4) |

7. Secondary Outcome: Change in Peak Force
Description: Change in peak force (N) during the 250 foot level propulsion task. Measurement was done using the SmartWheel.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit. There were technical issues preventing the SmartWheel data collection for 3 subjects in the intervention group
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 2 | 0
Newtons | 10.1 (14.4) |

8. Secondary Outcome: Change in Mechanical Effective Force
Description: Change in mechanical effective force during 250 foot level propulsion task (no unit) Measurement will be done using the SmartWheel.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit. There were technical issues prevention SmartWheel data collection for 3 subjects in the intervention group.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 2 | 0
unitless | 0.06 (0.17) |

9. Secondary Outcome: Wheelchair Transfer Ability
Description: Measurement of relative transfer range. Measured as the change in relative uphill (maximum) transfer height (inches).
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit
Measure: Median (Full Range); unit: inches
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 5 | 0
inches | 1 [-2 to 3] |

10. Secondary Outcome: Power Output
Description: Measurement of peak power output (watts/kg) using the Load Arm Ergometer.
Time Frame: Baseline and 12 weeks
Population: Subjects in the control group withdrew before the 12 week visit
Measure: Mean (Standard Deviation); unit: Watts/kg
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
Number analyzed (Participants) | 5 | 0
Watts/kg | 0.5 (1.5) |

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | Resistance Training - Vibrating Dumbbell | Resistance Training - Standard Dumbbell
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02998021/Prot_SAP_000.pdf